CLINICAL TRIAL: NCT06540807
Title: SafeHeal Anastomosis Feasibility Evaluation (SAFE)-2023 Study: A Study to Investigate the Performance and Safety of the Colovac 2 Colorectal Anastomosis Protection Device
Brief Title: SafeHeal Anastomosis Feasibility Evaluation (SAFE)-2023 Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SafeHeal Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAFE-2023
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Colovac (Experimental): The Colovac device will be implanted for approximately 10 days.
  Interventions: Device: Colovac Colorectal Anastomosis Protection Device; Procedure: Stoma creation

INTERVENTIONS:
Device: Colovac Colorectal Anastomosis Protection Device — A removable, temporary intraluminal bypass device designed to safely postpone the creation of a protective stoma until 10 days after surgery for only patients who need it (do not have a healed anastomosis)
  Other Names: Colovac 2
Procedure: Stoma creation — Diverting loop ileostomy

SUMMARY:
A feasibility study to assess the early safety and effectiveness of the Colovac 2 device in providing temporary protection of the anastomosis in patients undergoing low anterior resection for colon cancer.

DETAILED DESCRIPTION:
A primary diverting stoma is widely used by surgeons to bypass the low rectal anastomosis and reduce morbidity associated with anastomotic leaks. Typically, a stoma is created for all high-risk patients which means that many patients are exposed to potentially serious complications associated with the stoma itself without any clinical benefit.

Colovac is a local, temporary, minimally invasive bypass device that protects the anastomosis and safely postpones stoma creation for 10 days after surgery. By postponing stoma creation for 10 days, Colovac allows stoma avoidance in all patients except those whose anastomosis have not healed by 10 days after surgery, allowing the others to return to normal activity more quickly and safely.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Eligible to undergo open or minimally invasive sphincter-sparing low anterior resection with planned diverting loop ileostomy for malignancy, based on multidisciplinary team recommendations
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2History of left sided colitis
* Willingness to comply with protocol-specific treatment and study visits and to sign a written Informed Consent Form

Exclusion Criteria:

* History of left sided colitis
* Known allergy to nickel or other components of the Colovac 2 System
* Pregnant or nursing female subject
* Concomitant major surgical procedure in combination with Colorectal resection (i.e., hepatectomy)
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation, impair the ability of the participant to undergo protocol described procedures or interfere with the interpretation of study results including, but not limited to:
* Stage IV colorectal cancer unless curative intent R0 resection is planned AND there is no associated peritoneal disease
* Immunodeficiency (CD4+ count < 500 CU MM)
* Systemic steroid therapy within the past 6 months
* Systemic infection at the time of surgery or requiring systemic antimicrobial therapy up to 1 week before surgery
* Major surgical or interventional procedures within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study
* Diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, intraabdominal infection, ischemic bowel, carcinomatosis
* Fecal incontinence, involvement of sphincter by the neoplastic disease or evidence of extensive local disease in the pelvis seen on pre-operative imaging
* Severe malnutrition which is defined as at least 10% weight loss within 3 months prior to enrollment.
* Occurrence of any of the following during the colorectal surgery:

  1. Blood loss (>750 cc)
  2. Blood transfusion
  3. Any new sign of ischemia
  4. Positive air leak test
  5. Inadequate bowel preparation
  6. Anastomosis location greater than 15 cm from the anal verge
  7. Other intra-operative risks that preclude the subject from undergoing the procedure with the investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Migration | 10 days
  Rate of clinically significant device migration The rate of subjects for which the device has migrated clinically significant during its 10-day implant period.

CONTACTS AND LOCATIONS:
Overall Officials: Okiljon Rahimov, MD, Principal Investigator — Republican Specialized Scientific and Practical Medical Center of Oncology and Radiology MoH of RUz; Narxodja Sametdinov, MD, Principal Investigator — Akfa Medline LLC
Locations (1):
- AKFA, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No